CLINICAL TRIAL: NCT01679639
Title: An Open-label, Fixed-sequence, Three-period, Single Group Study to Investigate the Effects of Rifampicin as an OATP1B1 Inhibitor and a CYP2C8 Inducer on the Pharmacokinetics of Aleglitazar in Healthy Subjects
Brief Title: A Study to Investigate the Effects of Rifampicin on the Pharmacokinetics of Aleglitazar in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: BP25561; 2012-002274-31 (EudraCT Number)
Record Dates: First submitted 2012-09-01; First posted 2012-09-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — aleglitazar; Rifampin

ARMS (1):
- Aleglitazar (Experimental)
  Interventions: Drug: aleglitazar; Drug: rifampicin

INTERVENTIONS:
Drug: aleglitazar — Single dose of aleglitazar in Periods 1, 2, 3
Drug: rifampicin — Single dose in Periods 1 and 2; multiple doses in Period 3

SUMMARY:
This open-label, fixed-sequence, three-period, single group study will evaluate the effects of rifampicin on the pharmacokinetics of aleglitazar in healthy volunteers. Volunteers will receive single doses of aleglitazar in all three periods and single doses of rifampicin in periods 1 and 2, and multiple doses in period 3. The anticipated time on study treatment is up to 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, aged 18 to 55 years inclusive at the time of screening
* Body mass index (BMI) between 18.0 and 35.0 kg/m2 inclusive
* Females must be surgically sterile or use two acceptable methods of contraception
* Non-smoker or currently smoking less than five cigarettes/day and willing to abstain from smoking during the study

Exclusion Criteria:

* Any clinically relevant abnormal laboratory test results at screening or on Day -1 of all periods, as judged by the Investigator
* A history of clinically significant disorders (e.g., gastro-intestinal, cardiovascular, hepatic)
* Infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* An average alcohol intake of more than 14 units per week
* Volunteers diagnosed, or suspected of having porphyria, and subjects with first degree relatives diagnosed, or suspected of having porphyria
* Diagnosis of Gilberts Syndrome
* A positive screen for drugs of abuse at screening or on admission to the clinical unit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the plasma concentration time curve | Period 1 and 2: Predose and days 1 to 5; Period 3: Days 5 to 12

SECONDARY OUTCOMES:
Safety: incidence of adverse events | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Manchester, United Kingdom